CLINICAL TRIAL: NCT01602354
Title: Endotoxin Activity Assay as a Prognostic Factor in Gram-negative Septic Shock
Brief Title: Endotoxin in Gram-negative Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Imma Tatiana Borrelli, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: EAA G- SEP
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Gram Negative Septic Shock
Keywords: Endotoxin Activity Assay; Gram negative; Septic Shock; EAA
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gram-negative Septic shock: Patients affected by Gram-negative septic shock

SUMMARY:
The purpose of this observational study is to determine whether endotoxin levels and/or their trends can be considered predictive of morbility or mortality in septic shock caused by gram-negative bacteria, searching also for a possible correlation with Simplified Acute Physiology Score (SAPS II), Sequential Organ Failure Assessment (SOFA), White Blood Cells (WBC) and Platelets (PLT).

DETAILED DESCRIPTION:
Medical literature states that Endotoxin (a structural molecule of the Gram-negative bacteria extracellular membrane) is able to activate target cells such as macrophages and neutrophils, inducing them to produce and release cytokine, nitric oxide and other mediators that cause a systemic inflammatory response that can evolve until to endothelial damage, shock and multi-organ failure (MOF).

Since 2004 it has been possible to better determine the concentration and the activity of endotoxin in plasma, thanks to a reliable and quick to implement method: the EAA (Endotoxin Activity Assay) test, which is an alternative technique for detecting endotoxin in whole blood based on the detection of enhanced respiratory burst activity in neutrophils following their priming by complexes of endotoxin and a specific anti-endotoxin antibody. The EAA shows excellent performance characteristics in recovering endotoxin from spiked samples and can be performed within 30 min, using less than 100µl whole blood.

Participants of this study (all affected by gram-negative septic shock) will show different values of endotoxin in their blood samples during their stay in Intensive Care Unit (ICU), and the investigators will try to figure out if these values and their trends can be somehow predictive of morbility and/or mortality, despite the small number of septic patients and the heterogeneity of their clinical picture.

So, if endotoxin induces sepsis, can the investigators also state that high values and/or trends of endotoxin can be correlated to severity of disease?

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe sepsis or septic shock
* acquisition of informed consent
* age over 18 years old

Exclusion Criteria:

* any diagnosis different from severe sepsis or septic shock
* rejection of informed consent by participant
* age under 18 years old
* any clinic condition considered not suitable by researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care Unit with a diagnosis of severe sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Level of Endotoxin in blood samples | admission date (baseline)
  Values of endotoxin are also compared to SOFA, SAPSII, PLT, WBC
Change of Endotoxin from baseline | 3 days after admission
  Values of endotoxin are also compared to SOFA, SAPSII, PLT, WBC
Change of Endotoxin from baseline | 7 dayf after admission
  Values of endotoxin are also compared to SOFA, SAPSII, PLT, WBC

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Forfori, Researcher, Study Director — Department of Intensive Care Unit, Azienda Ospedaliero-Universitaria (AOU) Pisana; Francesco Giunta, Professor, Study Chair — Depatment of Intensive Care Unit, AOU Pisana; Imma Tatiana Borrelli, Doctor, Principal Investigator — Department of Intensive Care Unit, AOU Pisana
Locations (1):
- Department of Intensive Care Unit, AOU Pisana, Pisa, Italy